CLINICAL TRIAL: NCT04965727
Title: Deep Brain Stimulation of the Lateral Hypothalamus to Augment Motor Function of Patients With Spinal Cord Injury
Acronym: HoT-DBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jocelyne Bloch (Other)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Sponsor-Investigator, Jocelyne Bloch, Professor, Neurosurgeon, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HoT-DBS2021
Record Dates: First submitted 2021-05-31; First posted 2021-07-16 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Deep Brain Stimulation; Neuro: Spinal Cord Injury
Keywords: SCI; DBS; Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Single site, interventional, non-randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep brain stimulation (Experimental): Participants will undergo a surgery for Deep Brain Stimulation (DBS). The neurostimulation system will be used for neuro-rehabilitation of the motor function.
  Participants will follow a 3-month neuro-rehabilitation using DBS at a frequency of 3 times per week with physiotherapist.
  Interventions: Procedure: Device implantation

INTERVENTIONS:
Procedure: Device implantation — The intervention involves the insertion of lead electrodes (Medtronic SenSight Directional Lead) in the right and left lateral hypothalamus through craniotomy and an implantable pulse generator (Medtronic Model B35200 Percept™ PC) in the upper part of the pectoralis major (under the clavicle).

SUMMARY:
The purpose of this study is to evaluate safety of Deep Brain Stimulation (DBS) of the lateral hypothalamus (LH) and whether the use of DBS can increase motor performance in patients with chronic spinal cord injury (SCI). The hypothesis, based on preclinical findings, is that DBS of the lateral hypothalamus can acutely augment leg motor function after SCI, and that the use of lateral hypothalamus DBS can be an adjunct during rehabilitation to promote recovery and long-term neuroplasticity.

DETAILED DESCRIPTION:
The investigators hypothesize that deep brain stimulation (DBS) delivered in the lateral hypothalamus (LH) can augment leg motor function in humans with SCI. DBS is a well-established neurosurgical technique that is used routinely in humans. For example, DBS is commonly used to regulate the activity of basal ganglia circuits in order to treat movement disorders like Parkinson's disease or tremor. For the past decade, the hypothalamus has been safely targeted to treat diseases such as obesity and cluster headache.

In this study, The investigators propose to test the safety and preliminary efficacy of Lateral Hypothalamus DBS in 3 individuals with incomplete SCI, as a potential basis for larger clinical trials. The investigators anticipate that such clinical trials will evaluate the respective impact of, and potential synergy between, DBS of the lateral hypothalamus and epidural electrical stimulation of the lumbar spinal cord to augment recovery from SCI.

The study intervention consists of 7 phases preceded by pre-screening:

* Screening and enrolment
* Baseline - Pre-implantation
* Surgery
* Calibration
* Pre-rehabilitation
* Rehabilitation
* Post-rehabilitation
* (Optional and conditional): safety follow-up period

Measures will be performed before surgical intervention, after surgery but before training (Pre-rehabilitation), at regular intervals during training and at the end of the training phase (post-rehabilitation).

The study will take place at the CHUV (Lausanne, Switzerland). A total of 3 participants will be enrolled in the study and implanted with the Medtronic Percept PC and 2 Medtronic SenSight DIrectional lead (left and right LH). All participants will undergo the same treatment and procedures. The active duration of the study will be approximately 7 to 8 months.

If deemed safe and beneficial by the Principal Investigator, participants may keep using the investigational device independently for 3 more years by entering the safety follow-up period at the end of the main study phase.

ELIGIBILITY:
Inclusion Criteria:

* SCI graded as American Spinal Injury Association Impairment Scale (AIS) C or D (able to walk independently for a few meters with a walker)
* Focal spinal cord disorder caused by trauma
* Minimum 12 months post-injury
* Stable medical, physical and psychological condition as considered by Investigators
* Able to understand and interact with the study team in French or English
* Adequate care-giver support and access to appropriate medical care in patient's home community
* Must agree to comply in good faith with all conditions of the study and to attend all required study training and visit
* Must provide and sign Informed Consent prior to any study related procedures

Exclusion Criteria:

* Limitation of walking function based on accompanying (CNS) disorders (i.e., systemic malignant disorders, cardiovascular disorders restricting physical training, peripheral nerve disorders)
* History of significant autonomic dysreflexia
* Cognitive/brain damage
* Epilepsy
* Use of an intrathecal baclofen pump
* Any active implanted cardiac device such as pacemaker or defibrillator
* Any indication that would require diathermy
* Increased risk for defibrillation
* Severe joint contractures disabling or restricting lower limb movements
* Hematological disorders with increased risk for surgical interventions
* Congenital or acquired lower limb abnormalities (affection of joints and bone)
* Women who are pregnant (pregnancy test obligatory for woman of childbearing potential) or breastfeeding
* Lack of safe contraception for women of childbearing capacity
* Spinal cord lesion due to either a neurodegenerative disease or a tumor
* Gastrointestinal ulcers in the last five years
* Known or suspected eye disorders or diseases
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.)
* Any other anatomic or co-morbid conditions that, in the Investigator's opinion, could limit the patient's ability to participate in the study or to comply with follow-up requirements, or impact the scientific soundness of the study results
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Participation in another locomotor training study
* Refusal to be informed of any finding during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Occurence of all SAEs and AEs that are deemed related or possibly related to study procedure or to study investigational system, from implantation up to the end of the study | Through study completion, an average of 6 months
  Evaluate the safety of the approach in terms of tolerability of deep brain stimulation of the lateral hypothalamus in patients with chronic spinal cord injury (> 1 year)

SECONDARY OUTCOMES:
Lower Extremity Motor Strength (M0-M5 score according to the AIS scale) | Baseline ; pre-rehabilitation (2-3 weeks after surgery) ; after 1 month of rehabilitation ; after 3 months of rehabilitation
  The American Spinal Injury Association (ASIA) Standard Neurological CLassification of Spinal Cord Injury is a standard method of assessing the neuological status, including motor and sensory evaluations, of a person who has sustained a spinal cord injury
Walking Index for Spinal Cord Injury (WISCI II) | Baseline ; pre-rehabilitation (2-3 weeks after surgery) ; after 1 month of rehabilitation ; after 3 months of rehabilitation
  The WISCI II is an ordinal scale to assess walking function
Walking speed (10MWT/6MWT) | Baseline ; pre-rehabilitation (2-3 weeks after surgery) ; after 1 month of rehabilitation ; after 3 months of rehabilitation
  10 meter walk test (10MWT) and 6 minutes walk test (6MWT) are common tests used to measure walking speed and lomotor performance

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Bloch, MD, Principal Investigator — CHUV
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angeli CA, Boakye M, Morton RA, Vogt J, Benton K, Chen Y, Ferreira CK, Harkema SJ. Recovery of Over-Ground Walking after Chronic Motor Complete Spinal Cord Injury. N Engl J Med. 2018 Sep 27;379(13):1244-1250. doi: 10.1056/NEJMoa1803588. Epub 2018 Sep 24. PMID 30247091
- [Background] Gill ML, Grahn PJ, Calvert JS, Linde MB, Lavrov IA, Strommen JA, Beck LA, Sayenko DG, Van Straaten MG, Drubach DI, Veith DD, Thoreson AR, Lopez C, Gerasimenko YP, Edgerton VR, Lee KH, Zhao KD. Neuromodulation of lumbosacral spinal networks enables independent stepping after complete paraplegia. Nat Med. 2018 Nov;24(11):1677-1682. doi: 10.1038/s41591-018-0175-7. Epub 2018 Sep 24. PMID 30250140
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Hou JM, Sun TS, Xiang ZM, Zhang JZ, Zhang ZC, Zhao M, Zhong JF, Liu J, Zhang H, Liu HL, Yan RB, Li HT. Alterations of resting-state regional and network-level neural function after acute spinal cord injury. Neuroscience. 2014 Sep 26;277:446-54. doi: 10.1016/j.neuroscience.2014.07.045. Epub 2014 Jul 30. PMID 25086312
- [Background] Cortes M, Medeiros AH, Gandhi A, Lee P, Krebs HI, Thickbroom G, Edwards D. Improved grasp function with transcranial direct current stimulation in chronic spinal cord injury. NeuroRehabilitation. 2017;41(1):51-59. doi: 10.3233/NRE-171456. PMID 28505987
- [Background] Kumru H, Benito-Penalva J, Valls-Sole J, Murillo N, Tormos JM, Flores C, Vidal J. Placebo-controlled study of rTMS combined with Lokomat(R) gait training for treatment in subjects with motor incomplete spinal cord injury. Exp Brain Res. 2016 Dec;234(12):3447-3455. doi: 10.1007/s00221-016-4739-9. Epub 2016 Jul 28. PMID 27469242
- [Background] Kim LH, Sharma S, Sharples SA, Mayr KA, Kwok CHT, Whelan PJ. Integration of Descending Command Systems for the Generation of Context-Specific Locomotor Behaviors. Front Neurosci. 2017 Oct 18;11:581. doi: 10.3389/fnins.2017.00581. eCollection 2017. PMID 29093660
- [Background] van den Brand R, Heutschi J, Barraud Q, DiGiovanna J, Bartholdi K, Huerlimann M, Friedli L, Vollenweider I, Moraud EM, Duis S, Dominici N, Micera S, Musienko P, Courtine G. Restoring voluntary control of locomotion after paralyzing spinal cord injury. Science. 2012 Jun 1;336(6085):1182-5. doi: 10.1126/science.1217416. PMID 22654062
- [Background] Sinnamon HM. Locomotor stepping elicited by electrical stimulation of the hypothalamus persists after lesion of descending fibers of passage. Physiol Behav. 1990 Aug;48(2):261-6. doi: 10.1016/0031-9384(90)90310-z. PMID 2255729
- [Background] Sinnamon HM. Preoptic and hypothalamic neurons and the initiation of locomotion in the anesthetized rat. Prog Neurobiol. 1993 Sep;41(3):323-44. doi: 10.1016/0301-0082(93)90003-b. PMID 8105509